CLINICAL TRIAL: NCT01155479
Title: A Phase 3, Double-Blind, Double-Dummy, Placebo- and Active-Controlled Dose-Range-Finding Efficacy and Safety Study of Preladenant in Subjects With Early Parkinson's Disease
Brief Title: A Placebo- and Active-Controlled Study of Preladenant in Early Parkinson's Disease (PD) (P05664)
Acronym: PARADYSE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termininated for business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05664; 2009-013552-72 (EudraCT Number); MK-3814-024 (Other: Merck Study Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Tablets; rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Preladenant 2 mg (Experimental): Preladenant 2 mg oral tablet and placebo for rasagiline taken in the morning (AM) followed by preladenant 2 mg oral tablet taken in the evening (PM) for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
  Interventions: Drug: Preladenant 2 mg tablet; Drug: Placebo for Rasagiline 1 mg capsule
- Preladenant 5 mg (Experimental): Preladenant 5 mg oral tablet and placebo for rasagiline taken in the AM followed by preladenant 5 mg taken in the PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
  Interventions: Drug: Preladenant 5 mg tablet; Drug: Placebo for Rasagiline 1 mg capsule
- Preladenant 10 mg (Experimental): Preladenant 10 mg oral tablet and placebo for rasagiline taken in the AM followed by preladenant 10 mg taken in the PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
  Interventions: Drug: Preladenant 10 mg tablet; Drug: Placebo for Rasagiline 1 mg capsule
- Placebo (Placebo Comparator): Placebo for preladenant and placebo for rasagiline taken in the AM followed by placebo for preladenant taken in the PM for 26 weeks (Part 1); preladenant 5 mg was taken twice daily for 26 weeks (Part 2).
  Interventions: Drug: Preladenant 5 mg tablet; Drug: Placebo for Rasagiline 1 mg capsule; Drug: Placebo for Preladenant
- Rasagiline (Active Comparator): Rasagiline 1 mg oral capsule and placebo for preladenant taken in the AM followed by placebo for preladenant taken in the PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
  Interventions: Drug: Rasagiline 1 mg capsule; Drug: Placebo for Preladenant

INTERVENTIONS:
Drug: Preladenant 2 mg tablet — Preladenant 2 mg oral tablet taken twice daily
  Other Names: SCH 420814
  Arms: Preladenant 2 mg
Drug: Preladenant 5 mg tablet — Preladenant 5 mg oral tablet taken twice daily
  Other Names: SCH 420814
  Arms: Placebo; Preladenant 5 mg
Drug: Preladenant 10 mg tablet — Preladenant 10 mg oral tablet taken twice daily
  Other Names: SCH 420814
  Arms: Preladenant 10 mg
Drug: Rasagiline 1 mg capsule — Rasagiline 1 mg oral capsule taken once daily
  Other Names: Azilect
  Arms: Rasagiline
Drug: Placebo for Rasagiline 1 mg capsule — Placebo for rasagiline 1 mg oral capsule taken once daily
  Arms: Placebo; Preladenant 10 mg; Preladenant 2 mg; Preladenant 5 mg
Drug: Placebo for Preladenant — Placebo for preladenant 2 mg, 5 mg, or 10 mg oral tablet taken twice daily
  Arms: Placebo; Rasagiline

SUMMARY:
This is a one year, 2-part study to determine the efficacy and safety of preladenant, an adenosine type 2a (A2a) receptor antagonist. The purpose of Part 1 (first 26 weeks) is to determine if preladenant is effective in the treatment of early Parkinson's Disease. The purpose of Part 2 (second 26 weeks) is to determine if preladenant is safe and well tolerated. The primary efficacy hypothesis is that at least the 10 mg twice daily dose of preladenant is superior to placebo as measured by the change from Baseline to Week 26 in the sum of Unified Parkinson's Disease Rating Scale (UPDRS) Parts 2 and 3 scores (UPDRS2+3).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of idiopathic PD for < 5 years.
* If receiving amantadine and/or anticholinergics, must have been on a stable regimen of treatment for at least the 5 weeks immediately before Screening. (Note: Participants who are not taking any medications for PD are permitted to enroll in this trial.)
* Must have a UPDRS Part 3 score of ≥10, a Hoehn and Yahr Stage ≤3, be ≥30 to ≤85 years of age, and have results of Screening clinical laboratory tests drawn within 5 weeks prior to randomization, clinically acceptable to the investigator, and not within the parameters specified for exclusion.
* If sexually active or plan to be sexually active, must agree to use a highly effective method of birth control while the participant is in the study and for 2 weeks after the last dose of study drug. A male participant must also not donate sperm during the trial and within 2 weeks after the last dose of study drug.

Exclusion Criteria:

* Must not have a form of drug-induced or atypical Parkinsonism, cognitive impairment (ie, Montreal Cognitive Assessment [MoCA] score <22), bipolar disorder, untreated major depressive disorder, schizophrenia, or other psychotic disorder; history of exposure to a known neurotoxin, or any neurological features not consistent with the diagnosis of PD as assessed by the investigator.
* Must not have had surgery for PD.
* Must not have a history of repeated strokes with stepwise progression of Parkinsonism or head injuries, or a stroke within 6 months of screening; poorly controlled diabetes; abnormal renal function; or a severe or ongoing unstable medical condition.
* Must not have failed to show a therapeutic response if a diagnostic levodopa (L dopa) challenge had been done with a large test dose (>500 mg) of L dopa (if malabsorption excluded), or failed to respond to an adequate previous treatment with dopaminergic therapy.
* Must not have been treated with L dopa or dopamine agonists for 30 days or more. A participant who has been treated with L-dopa or dopamine agonists for <30 days will be allowed to enter the study. These participants must stop taking dopaminergic medication 30 days prior to Randomization.
* Must not be at imminent risk of self-harm or harm to others.
* Must not have elevated blood pressure (BP) (systolic BP ≥150 mm Hg or diastolic BP ≥95 mm Hg) that cannot be adequately controlled with antihypertensive medication, as demonstrated by 2 BP measurements meeting acceptable BP criterion at consecutive scheduled or unscheduled visits between Screening and Randomization (a 5-6 week period), one of which must be the Randomization visit.
* Must not have had any clinically significant cardiovascular event or procedure for 6 months prior to Randomization, including, but not limited to, myocardial infarction, angioplasty, unstable angina, or heart failure; and a participant must not have heart failure staged New York Heart Association Class III or IV.
* Must not have an alanine aminotransferase (ALT) or aspartate amino transferase (AST) ≥ 3 x the upper limit of normal (ULN) or total bilirubin (T BIL) ≥ 1.5 x ULN.
* Must not have active serologically-confirmed hepatic dysfunction (defined as viral infection [Hepatitis B, C, or E; Epstein-Barr virus (EBV)]; cytomegalovirus [CMV] or a history of diagnosis of drug- or alcohol-induced hepatic toxicity or frank hepatitis, or a history of diagnosis of drug- or alcohol-induced hepatic toxicity or frank hepatitis.)
* Must not have a history within the past 5 years of a primary or recurrent malignant disease with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with a normal prostate-specific antigen (PSA) post resection.
* Must not have received certain prespecified medications or ingested high tyramine-containing aged cheeses (eg, Stilton) for a prespecified time window before the trial, during the trial, and for 2 weeks after the trial.
* Must not have an average daily consumption of more than three 4 ounce glasses (118 mL) of wine or the equivalent.
* Must not have a severe or ongoing unstable medical condition (eg, any form of clinically significant cardiac disease, symptomatic orthostatic hypotension, seizures, or alcohol/drug dependence.)
* Must not have allergy/sensitivity to investigational product(s) or its/their excipients.
* Must not be breast-feeding, considering breast-feeding, pregnant or intending to become pregnant.
* Must not have used preladenant ever, or any investigational drugs within 90 days immediately before screening.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2010-07-06 (Actual); Primary Completion 2013-07-16 (Actual); Study Completion 2013-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Stocchi F, Rascol O, Hauser RA, Huyck S, Tzontcheva A, Capece R, Ho TW, Sklar P, Lines C, Michelson D, Hewitt DJ; Preladenant Early Parkinson Disease Study Group. Randomized trial of preladenant, given as monotherapy, in patients with early Parkinson disease. Neurology. 2017 Jun 6;88(23):2198-2206. doi: 10.1212/WNL.0000000000004003. Epub 2017 May 10. PMID 28490648
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05664&kw=P05664&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of idiopathic PD for less than 5 years were selected to participate in this study.
Pre-assignment Details: In Part 1, participants were randomized to one of five treatment groups and treated for 26 weeks. In Part 2, which was conducted for an additional 26 weeks, participants continued taking the same study treatment from Part 1, except for placebo participants who were re-assigned to receive preladenant 5 mg twice daily.
Groups:
- Preladenant 2 mg: Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
- Preladenant 5 mg: Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
- Preladenant 10 mg: Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
- Placebo: Participants received placebo for preladenant and placebo for rasagiline in the AM followed by placebo for preladenant in the PM for 26 weeks (Part 1); preladenant 5 mg was taken twice daily for 26 weeks (Part 2).
- Rasagiline: Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
Period: Part I
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline
Started | 204 | 204 | 206 | 204 | 204
Treated | 200 | 202 | 204 | 198 | 203
Completed | 166 | 177 | 167 | 177 | 181
Not Completed | 38 | 27 | 39 | 27 | 23
Not completed — Adverse Event | 13 | 8 | 18 | 7 | 6
Not completed — Administrative | 2 | 2 | 2 | 0 | 0
Not completed — Did Not Meet Protocol Eligibility | 3 | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 11 | 13 | 8 | 8 | 9
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Treatment Failure | 3 | 0 | 3 | 1 | 2
Not completed — Did Not Receive Treatment | 4 | 2 | 2 | 6 | 1
Not completed — Non-Compliance with Protocol | 2 | 1 | 3 | 3 | 2
Period: Part II
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline
Started | 166 | 177 | 167 | 177 | 181
Completed | 107 | 116 | 109 | 127 | 126
Not Completed | 59 | 61 | 58 | 50 | 55
Not completed — Adverse Event | 7 | 6 | 8 | 3 | 4
Not completed — Administrative | 43 | 49 | 36 | 38 | 46
Not completed — Withdrawal by Subject | 8 | 4 | 12 | 7 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Treatment Failure | 0 | 1 | 2 | 0 | 1
Not completed — Non-Compliance with Protocol | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All Participants as Randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline | Total
Number analyzed (Participants) | 204 | 204 | 206 | 204 | 204 | 1022
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (10.5) | 62.3 (10.2) | 63.8 (11.1) | 63.3 (10.0) | 62.9 (10.2) | 63.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 90 | 90 | 82 | 85 | 425
  Male | 126 | 114 | 116 | 122 | 119 | 597

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Sum of Unified Parkinson's Disease Rating Scale Parts 2 and 3 Scores (UPDRS2+3)
Description: The UPDRS is a clinician based rating scale used to measure motor impairments and disability. The UPDRS assesses six features of PD impairment. These are evaluated using a combination of data collected by interview and examination of the participant. The UPDRS Part 2 is the Activities of Daily Living (ADL) score and can range from 0-52 as determined by the physician. The UPDRS Part 3 is the Motor Examination (Total Motor Score [TMS]) and is defined as the total score, ranging from 0-108 as determined by the physician, of the tests given in the motor examination section. The combined scores of Parts 2 and 3 can range from 0-160 with the higher score indicating the worse condition. Change from baseline was analyzed using a constrained longitudinal analysis (cLDA) model with treatment, time, strata and treatment-by-time interaction as fixed effects and participant as a random effect.
Time Frame: Baseline and Week 26
Population: Full Analysis Set (FAS): All randomized and treated participants with at least one post-baseline value.
Measure: Mean (Standard Error); unit: Score on a Scale
Groups:
- Preladenant 2 mg (Part 1): Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks.
- Preladenant 5 mg (Part 1): Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks.
- Preladenant 10 mg (Part 1): Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks.
- Placebo (Part 1): Participants received placebo for preladenant and placebo for rasagiline in the AM followed by placebo for preladenant in the PM for 26 weeks.
- Rasagiline (Part 1): Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks.
Arm/Group | Preladenant 2 mg (Part 1) | Preladenant 5 mg (Part 1) | Preladenant 10 mg (Part 1) | Placebo (Part 1) | Rasagiline (Part 1)
Number analyzed (Participants) | 195 | 202 | 200 | 195 | 195
Score on a Scale | 0.3 (0.63) | -1.0 (0.60) | -1.8 (0.61) | -2.2 (0.61) | -1.9 (0.61)
Statistical Analysis 1: Comparison: Preladenant 2 mg (Part 1) vs Placebo (Part 1); Preladenant 2 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.0033, constrained longitudinal analysis; Difference in Estimated Means = 2.60, 95% CI 2-sided [0.86 to 4.30]
Statistical Analysis 2: Comparison: Preladenant 5 mg (Part 1) vs Placebo (Part 1); Preladenant 5 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.1382, constrained longitudinal analysis; Difference in Estimated Means = 1.30, 95% CI 2-sided [-0.41 to 2.94]
Statistical Analysis 3: Comparison: Preladenant 10 mg (Part 1) vs Placebo (Part 1); Preladenant 10 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.6378, constrained longitudinal analysis; Difference in Estimated Means = 0.40, 95% CI 2-sided [-1.29 to 2.11]
Statistical Analysis 4: Comparison: Placebo (Part 1) vs Rasagiline (Part 1); Rasagiline (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.6923, constrained longitudinal analysis; Difference in Estimated Means = 0.30, 95% CI 2-sided [-1.35 to 2.03]

2. Secondary Outcome: Percentage of Responders (Participants With a ≥20% Improvement in UPDRS2+3)
Description: UPDRS is a clinician based rating scale used to measure motor impairments and disability; it assesses 6 features of PD impairment. These are evaluated using a combination of data collected by interview and examination of the participant. UPDRS Part 2 is Activities of Daily Living score and ranges from 0-52. UPDRS Part 3 is Motor Examination and ranges from 0-108. The combined scores of Parts 2 and 3 can range from 0-160 with the higher score indicating the worse condition. A Responder is defined as a participant with at least 20% improvement in UPDRS2+3 from Baseline to Week 26 (End of Part 1 Treatment); a participant with at least a 20% decrease from Baseline score in UPDRS2+3 is defined as a responder. The proportion of Responders was analyzed using a generalized linear mixed model with treatment effect, strata and Baseline UPDRS2+3 as a covariate, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 26
Population: Full Analysis Set (FAS): All randomized and treated participants with at least one post-baseline value.
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Groups:
- Preladenant 2 mg (Part 1): Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks. The number of participants analyzed (195) represents the number of randomized and treated participants with at least one post-treatment value.
- Preladenant 5 mg (Part 1): Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks. The number of participants analyzed (202) represents the number of randomized and treated participants with at least one post-treatment value.
- Preladenant 10 mg (Part 1): Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks. The number of participants analyzed (200) represents the number of randomized and treated participants with at least one post-treatment value.
- Placebo (Part 1): Participants received placebo for preladenant and placebo for rasagiline in the AM followed by placebo for preladenant in the PM for 26 weeks. The number of participants analyzed (195) represents the number of randomized and treated participants with at least one post-treatment value.
- Rasagiline (Part 1): Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks. The number of participants analyzed (195) represents the number of randomized and treated participants with at least one post-treatment value.
Arm/Group | Preladenant 2 mg (Part 1) | Preladenant 5 mg (Part 1) | Preladenant 10 mg (Part 1) | Placebo (Part 1) | Rasagiline (Part 1)
Number analyzed (Participants) | 195 | 202 | 200 | 195 | 195
Percentage of Responders | 25.90 [18.95 to 34.33] | 29.50 [22.50 to 37.72] | 31.50 [24.06 to 40.02] | 35.20 [27.49 to 43.82] | 33.10 [25.60 to 41.51]
Statistical Analysis 1: Comparison: Preladenant 2 mg (Part 1) vs Placebo (Part 1); Preladenant 2 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.0785, generalized linear mixed model — p-value is for the estimated Odds Ratio based on a generalized linear mixed model with baseline UPDRS2+3 as a covariate and treatment-by-time interaction as fixed effect and participant as random effect; Difference vs Placebo (%) = -9.7, 95% CI 2-sided [-21.0 to 1.82]
Statistical Analysis 2: Comparison: Preladenant 5 mg (Part 1) vs Placebo (Part 1); Preladenant 5 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.2735, generalized linear mixed model — [p-value comment as in outcome 2, analysis 1]; Difference vs Placebo (%) = -6.3, 95% CI 2-sided [-17.6 to 5.05]
Statistical Analysis 3: Comparison: Preladenant 10 mg (Part 1) vs Placebo (Part 1); Preladenant 10 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.4823, generalized linear mixed model — [p-value comment as in outcome 2, analysis 1]; Difference vs Placebo (%) = -3.7, 95% CI 2-sided [-15.2 to 7.99]
Statistical Analysis 4: Comparison: Placebo (Part 1) vs Rasagiline (Part 1); Rasagiline (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.6827, generalized linear mixed model — [p-value comment as in outcome 2, analysis 1]; Difference vs Placebo (%) = -2.3, 95% CI 2-sided [-13.9 to 9.24]

3. Secondary Outcome: Change From Baseline in the UPDRS Part 2 Score (Activities of Daily Living [ADL])
Description: The UPDRS is a clinician based rating scale used to measure motor impairments and disability. The UPDRS assesses six features of PD impairment. These are evaluated using a combination of data collected by interview and examination of the participant. The UPDRS Part 2 is the Activities of Daily Living (ADL) score and can range from 0-52 as determined by the physician with the higher score indicating the worse condition. Change from baseline was analyzed using a cLDA model with treatment, time, strata and treatment-by-time interaction as fixed effects and participant as a random effect.
Time Frame: Baseline and Week 26
Population: Full Analysis Set (FAS): All randomized and treated participants with at least one post-baseline value.
Measure: Mean (Standard Error); unit: Score on a Scale
Groups:
- Rasagiline (Part 1): Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks (Part 1) and then for another 26 weeks (Part 2).
Arm/Group | Preladenant 2 mg (Part 1) | Preladenant 5 mg (Part 1) | Preladenant 10 mg (Part 1) | Placebo (Part 1) | Rasagiline (Part 1)
Number analyzed (Participants) | 195 | 202 | 200 | 195 | 195
Score on a Scale | 0.30 (0.22) | 0.10 (0.21) | -0.20 (0.21) | -0.40 (0.21) | -0.20 (0.21)
Statistical Analysis 1: Comparison: Preladenant 2 mg (Part 1) vs Placebo (Part 1); Preladenant 2 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.0235, constrained longitudinal analysis; Difference in Estimated Means = 0.70, 95% CI 2-sided [0.09 to 1.27]
Statistical Analysis 2: Comparison: Preladenant 5 mg (Part 1) vs Placebo (Part 1); Preladenant 5 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.1093, constrained longitudinal analysis; Difference in Estimated Means = 0.50, 95% CI 2-sided [-0.11 to 1.04]
Statistical Analysis 3: Comparison: Preladenant 10 mg (Part 1) vs Placebo (Part 1); Preladenant 10 mg (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.5756, constrained longitudinal analysis; Difference in Estimated Means = 0.20, 95% CI 2-sided [-0.42 to 0.75]
Statistical Analysis 4: Comparison: Placebo (Part 1) vs Rasagiline (Part 1); Rasagiline (Part 1) vs Placebo (Part 1); Test type: Superiority or Other; p = 0.6657, constrained longitudinal analysis; Difference in Estimated Means = 0.10, 95% CI 2-sided [-0.45 to 0.70]

4. Primary Outcome: Number of Participants With Adverse Events (AEs) in Part 1
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Day 1 to Week 26
Population: All Participants as Treated: All participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg (Part 1) | Preladenant 5 mg (Part 1) | Preladenant 10 mg (Part 1) | Placebo (Part 1) | Rasagiline (Part 1)
Number analyzed (Participants) | 200 | 202 | 204 | 198 | 203
Participants | 108 | 110 | 121 | 102 | 105

5. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE in Part 1
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Day 1 to Week 26
Population: All Participants as Treated: All participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg (Part 1) | Preladenant 5 mg (Part 1) | Preladenant 10 mg (Part 1) | Placebo (Part 1) | Rasagiline (Part 1)
Number analyzed (Participants) | 200 | 202 | 204 | 198 | 203
Participants | 13 | 8 | 20 | 8 | 6

6. Primary Outcome: Number of Participants With Adverse Events (AEs) in Part 2
Description: as for outcome 4
Time Frame: Week 27 to Week 52
Population: All Participants as Treated: All participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Groups:
- Preladenant 2 mg (Part 2): Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks.
- Preladenant 5 mg (Part 2): Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks.
- Preladenant 10 mg (Part 2): Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks.
- Placebo (Part 2): Participants who had received placebo to preladenant in Part 1 received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks.
- Rasagiline (Part 2): Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks.
Arm/Group | Preladenant 2 mg (Part 2) | Preladenant 5 mg (Part 2) | Preladenant 10 mg (Part 2) | Placebo (Part 2) | Rasagiline (Part 2)
Number analyzed (Participants) | 166 | 177 | 167 | 177 | 181
Participants | 116 | 120 | 113 | 120 | 119

7. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE in Part 2
Description: as for outcome 5
Time Frame: Week 27 to Week 52
Population: All Participants as Treated (APaT): All participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg (Part 2) | Preladenant 5 mg (Part 2) | Preladenant 10 mg (Part 2) | Placebo (Part 2) | Rasagiline (Part 2)
Number analyzed (Participants) | 166 | 177 | 167 | 177 | 181
Participants | 7 | 5 | 8 | 3 | 4

ADVERSE EVENTS:
Time Frame: Up to 54 weeks (including 2 weeks of follow-up)
Description: All Participants as Treated (APaT) - includes all participants who received at least one (1) dose of study drug.
Groups:
- Preladenant 2 mg - Part 1: Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks (Part 1).
- Preladenant 5 mg - Part 1: Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks (Part 1).
- Preladenant 10 mg - Part 1: Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks (Part 1).
- Placebo - Part 1: Participants received placebo for preladenant and placebo for rasagiline in the AM followed by placebo for preladenant in the PM for 26 weeks (Part 1).
- Rasagiline - Part 1: Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks (Part 1).
- Preladenant 2 mg - Part 2: Participants received preladenant 2 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 2 mg oral tablet in PM for 26 weeks (Part 2).
- Preladenant 5 mg - Part 2: Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg in the PM for 26 weeks (Part 2).
- Preladenant 10 mg - Part 2: Participants received preladenant 10 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 10 mg in the PM for 26 weeks (Part 2).
- Placebo/Preladenant 5 Mg-Part 2: Participants received preladenant 5 mg oral tablet and placebo for rasagiline in the AM followed by preladenant 5 mg oral tablet in the PM for 26 weeks (Part 2).
- Rasagiline - Part 2: Participants received rasagiline 1 mg oral capsule and placebo for preladenant in the AM followed by placebo for preladenant in PM for 26 weeks (Part 2).
Arm/Group | Preladenant 2 mg - Part 1 | Preladenant 5 mg - Part 1 | Preladenant 10 mg - Part 1 | Placebo - Part 1 | Rasagiline - Part 1 | Preladenant 2 mg - Part 2 | Preladenant 5 mg - Part 2 | Preladenant 10 mg - Part 2 | Placebo/Preladenant 5 Mg-Part 2 | Rasagiline - Part 2
Serious Adverse Events (participants affected / at risk) | 4/200 | 5/202 | 8/204 | 3/198 | 9/203 | 7/166 | 1/177 | 8/167 | 4/177 | 8/181
Other Adverse Events (participants affected / at risk) | 33/200 | 39/202 | 40/204 | 36/198 | 34/203 | 18/166 | 22/177 | 17/167 | 16/177 | 19/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg - Part 1 (N=200) | Preladenant 5 mg - Part 1 (N=202) | Preladenant 10 mg - Part 1 (N=204) | Placebo - Part 1 (N=198) | Rasagiline - Part 1 (N=203) | Preladenant 2 mg - Part 2 (N=166) | Preladenant 5 mg - Part 2 (N=177) | Preladenant 10 mg - Part 2 (N=167) | Placebo/Preladenant 5 Mg-Part 2 (N=177) | Rasagiline - Part 2 (N=181)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antinuclear Antibody Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinonasal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy of Partner (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden Cardiac Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg - Part 1 (N=200) | Preladenant 5 mg - Part 1 (N=202) | Preladenant 10 mg - Part 1 (N=204) | Placebo - Part 1 (N=198) | Rasagiline - Part 1 (N=203) | Preladenant 2 mg - Part 2 (N=166) | Preladenant 5 mg - Part 2 (N=177) | Preladenant 10 mg - Part 2 (N=167) | Placebo/Preladenant 5 Mg-Part 2 (N=177) | Rasagiline - Part 2 (N=181)
Constipation (Gastrointestinal disorders) | 5 (6) | 9 (10) | 11 (11) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 4 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (11) | 8 (8) | 6 (6) | 6 (6) | 3 (3) | 9 (9) | 3 (3) | 7 (8) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7) | 11 (12) | 5 (6) | 9 (9) | 10 (11) | 4 (4) | 1 (1) | 4 (4) | 1 (2) | 6 (7)
Headache (Nervous system disorders) | 13 (19) | 10 (13) | 15 (20) | 5 (7) | 10 (10) | 11 (16) | 4 (6) | 9 (11) | 5 (5) | 7 (8)
Tremor (Nervous system disorders) | 8 (15) | 7 (11) | 3 (3) | 11 (13) | 6 (8) | 7 (8) | 11 (12) | 5 (5) | 8 (10) | 6 (7)
Hypertension (Vascular disorders) | 4 (4) | 11 (13) | 11 (12) | 11 (12) | 11 (11) | 1 (1) | 5 (6) | 6 (7) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The Investigator further agrees to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment.